CLINICAL TRIAL: NCT02146001
Title: Reducing Sedentary Behavior vs. Increasing Physical Activity in Older Adults
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Bethany Barone Gibbs, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pitt Pepper 124078
Record Dates: First submitted 2014-03-03; First posted 2014-05-23 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Sedentary Lifestyle
Keywords: sedentary behavior; physical activity; older adults
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate-to-vigorous activity group (Active Comparator): This group will target achieving the current recommendations for physical activity in older adults. This is 150 minutes of moderate-to-vigorous activity per week.
  Interventions: Other: Moderate-to-vigorous activity group
- Reducing sedentary behavior group (Experimental): This group will target a 60 minute per day reduction in sedentary behavior using an objective activity monitor.
  Interventions: Other: Reducing sedentary behavior group

INTERVENTIONS:
Other: Reducing sedentary behavior group — This intervention will use individual counseling and the the BodyMedia armband to self-monitor sedentary behavior. The goal will be to decrease time spent in sedentary behavior by 60 minutes each day.
  Arms: Reducing sedentary behavior group
Other: Moderate-to-vigorous activity group — This group will be administered an individual, behavioral intervention using the BodyMedia armband to self-monitor physical activity. The prescription will be 150 minutes of moderate exercise (e.g. brisk walking) each week.
  Arms: Moderate-to-vigorous activity group

SUMMARY:
This study is a randomized trial that will compare the effects of two, 12-week activity interventions on patterns of physical activity, physical health, and quality of life measures in 40 older adults who are able to walk for exercise. One intervention will target 150 minutes per week of home-based moderate exercise (e.g. brisk walking), consistent with current recommendations. The other intervention will target a decrease in time spent in sedentary behaviors (e.g. sitting) of 60 minutes per day. Both interventions will wear an activity armband which will allow them to self-monitor their activity or sedentary behavior in real time using a smartphone. The armband will also provide objective data to an interventionist that will facilitate the intervention. The main outcome will be time spent in moderate exercise.

DETAILED DESCRIPTION:
Specific Aims: This application proposes to randomize community-dwelling, older adults to one of two, 12-week activity interventions that target either increased moderate-to-vigorous physical activity (MVPA) or decreased sedentary behavior (SED). The primary aim of this research is to evaluate the effect of a behavioral intervention targeting decreased SED vs. increased MVPA on objectively monitored activity (minutes of SED and MVPA). The secondary aim is to evaluate the effect of the SED intervention vs. the MVPA intervention on functional and psychosocial outcomes. To the investigators knowledge, this research will provide unique experimental evidence that SED can be altered in an older adult population and will yield key pilot data on the expected effect size for an intervention targeting SED vs. MVPA.

Background: The older adult population is the least active age group in the U.S. by two distinct metrics: a lack of MVPA and a high rate of SED (sitting without any significant exertion). This represents a public health opportunity because engaging in 150 minutes of MVPA is known to improve the risk of morbidity, mortality, and physical function. SED has emerged as a risk factor for adverse outcomes, independent of MVPA, and observational studies indicate that more SED is linked to an increased risk of clinical outcomes (mortality, diabetes, and cardiovascular disease) and worse aging outcomes, e.g. physical function. However, there exists no experimental data comparing interventions to reduce SED vs. increase MVPA in older adults.

Summary of Methods: The investigators propose a 2-arm randomized trial that will target increasing MVPA (Get Active) vs. decreasing SED (Sit Less) among community-dwelling, older adults from the Pepper Center Mobility Registry. The intervention will consist of a combination of in-person (Weeks 1-4, 6, 8, 10) and phone-based (Weeks 5, 7, 9, 11) individual counseling and will utilize the BodyMedia® Fit System (wearable armband with technology interface) to provide real-time feedback on daily MVPA or SED, which can be used by the subjects to self-monitor and by the interventionist to improve adherence. Assessments at baseline and 12 weeks will include objectively monitored minutes of MVPA and SED by a blinded armband, physical function (short physical performance battery, 400 meter walk, grip strength, gait speed), and assessment of subjective MVPA, SED, physical function, and psychosocial outcomes by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Currently engage in <60 minutes of MVPA per week
* Ability to complete a 400 meter walk test without an assistive device
* Access to a computer and compatible smartphone (Andriod or iPhone) for the use of the BodyMedia® Fit System to monitor Moderate -to - Vigorous physical activity or sedentary behavior
* Ability to provide medical clearance to participate in this study from their primary care physician

Exclusion Criteria:

* Unable to provide informed consent
* Household member on study staff
* Current or planned enrollment in another physical activity or weight loss program
* Cardiovascular event (heart attack, stroke, heart failure, revascularization procedure) in the last 6 months
* Current use of beta-blockers or other medication that could affect heart rate
* Currently treated for psychological issues, or taking psychotropic medications within the previous 6 months
* Comorbid condition that would limit participation in exercise (e.g. uncontrolled hypertension, severe arthritis, use of a assistive mobility device, currently undergoing treatment for cancer)
* >3 alcoholic beverages per day

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Barone Gibbs, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Physical Activity and Weight Management Research Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 241 subjects were screened. Of these 190 did not meet inclusion criteria, 13 declined to participate, and 38 were eligible and enrolled in the study.
Groups:
- Get Active: Targeting 150 minutes/week of moderate-to-vigorous intensity physical activity
- Sit Less: Targeting 1 hour less of sedentary time per day
Period: Overall Study
Arm/Group | Get Active | Sit Less
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Get Active | Sit Less | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (6.5) | 68.5 (6.5) | 67.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 14 | 18 | 32
  Non-white | 5 | 1 | 6
Body Mass Index, continuous [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (6.3) | 28.3 (4.8) | 28.6 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Objectively Monitored Sedentary Behavior
Description: Subjects will wear a BodyMedia SenseWearPro armband for 7 days during all waking hours at baseline and 12 weeks. This multi-sensor armband will give an estimate of time spent in sedentary behavior over a 1 week period. Sedentary time will be averaged across days and reported as hours per day.
Time Frame: Change from baseline to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: hours/day
Arm/Group | Get Active | Sit Less
Number analyzed (Participants) | 19 | 19
hours/day | -0.1 (0.4) | 0.6 (0.3)

2. Secondary Outcome: Change in Physical Function (Short Physical Performance Battery [SPPB])
Description: Physical function will be assessed by the Short Physical Performance Battery including a chair stand test (timed test to stand up and down 5 times without using hands), a 4-meter walk test for gait speed, and a standing balance test. Standard scoring of the SPPB was used where each test contributes up to 4 points x 3 tests and the score can, therefore, range from 0 (worst) to 12 (best).
Time Frame: Change from baseline to 12 weeks
Measure: Mean (Standard Error); unit: points
Arm/Group | Get Active | Sit Less
Number analyzed (Participants) | 19 | 19
points | 0.2 (0.2) | 0.5 (0.3)

3. Secondary Outcome: Change in Objectively-monitored Moderate-to-vigorous Physical Activity
Description: Subjects will wear a BodyMedia SenseWearPro armband for 7 days during all waking hours at baseline and 12 weeks (same as for the primary outcome of sedentary behavior). This multi-sensor armband will give an estimate of time spent in moderate-to-vigorous physical activity over a 1 week period.
Time Frame: Change from baseline to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: bouted minutes/week
Arm/Group | Get Active | Sit Less
Number analyzed (Participants) | 19 | 19
bouted minutes/week | 75 (22) | -7 (25)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Get Active | Sit Less
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No